CLINICAL TRIAL: NCT07313644
Title: Electrical Impedance Tomography-Guided Positive End-Expiratory Pressure Optimization in Patients With Trauma-Related and Postoperative Acute Respiratory Distress Syndrome
Brief Title: EIT-Guided PEEP Optimization in Trauma and Postoperative ARDS
Acronym: EIT-PEEP-SURG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nguyen Dang Thu (Other)
Collaborators: Hanoi Medical University (Other); Viet Duc University Hospital (Other)
Responsible Party: Sponsor-Investigator, Nguyen Dang Thu, Ph.D; M.D., Vietnam Military Medical University
Organization: Vietnam Military Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MinhGMHS 1879/GCN-HMUIRB
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Syndrome Distress; Positive End-Expiratory Pressure; Electrical Impedance Tomography; Trauma and Postoperative Pulmonary Insufficiency
Keywords: Acute respiratory syndrome distress; Positive End-Expiratory Pressure; electrical impedance tomography; Trauma and Postoperative; blood oxygenation; pulmonary mechanics
MeSH Terms: conditions — Respiratory Distress Syndrome; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Prospective, single center, ramdomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Device: electrical impedance tomography system (Enlight 2100, Timpel SA, Brazil).
  - Patients underwent airway suctioning and were deeply sedated (RASS ≤ -3) to abolish spontaneous breathing. PEEP titration was performed using an EIT system (Enlight 2100, Timpel SA, Brazil), with a silicone belt containing 32 surface electrodes positioned at the fourth to fifth intercostal space in accordance with the manufacturer's instructions.
  Pressure-controlled ventilation was applied with an inspiration pressure set at 15 cmH₂O and a set PEEP of 24 cmH₂O, with a maximum airway pressure limit of 40 cmH₂O. Ventilator settings were maintained for 30 seconds with an FiO₂ of 1.0. A decremental PEEP trial was then performed by reducing PEEP in 2 cmH₂O every 30 seconds until a PEEP of 6 cmH₂O was reached or the SpO₂ decreased to ≤ 80%.
  The EIT-guided optimal PEEP was defined as the PEEP level corresponding to the intersection point of the collapse and overdistension curves.
  Interventions: Device: EIT-giuded PEEP
- Control Group (Placebo Comparator): PEEP was set and adjusted according to the lower PEEP/FiO₂ table of the ARDS Network
  Interventions: Device: Control

INTERVENTIONS:
Device: EIT-giuded PEEP — Device: electrical impedance tomography system (Enlight 2100, Timpel SA, Brazil).
  - Patients underwent airway suctioning and were deeply sedated (RASS ≤ -3) to abolish spontaneous breathing. PEEP titration was performed using an EIT system (Enlight 2100, Timpel SA, Brazil), with a silicone belt containing 32 surface electrodes positioned at the fourth to fifth intercostal space in accordance with the manufacturer's instructions.
  Pressure-controlled ventilation was applied with an inspiration pressure set at 15 cmH₂O and a set PEEP of 24 cmH₂O, with a maximum airway pressure limit of 40 cmH₂O. Ventilator settings were maintained for 30 seconds with an FiO₂ of 1.0. A decremental PEEP trial was then performed by reducing PEEP in 2 cmH₂O every 30 seconds until a PEEP of 6 cmH₂O was reached or the SpO₂ decreased to ≤ 80%.
  The EIT-guided optimal PEEP was defined as the PEEP level corresponding to the intersection point of the collapse and overdistension curves.
  Arms: Intervention Group
Device: Control — PEEP was set and adjusted according to the lower PEEP/FiO₂ table of the ARDS Network
  Arms: Control Group

SUMMARY:
Acute respiratory distress syndrome (ARDS) remains a serious and often fatal complication in patients following severe trauma or major surgery. Mechanical ventilation is essential for supportive care in this population, but may aggravate lung injury when suboptimal ventilatory settings are applied. Positive end-expiratory pressure (PEEP) is crucial for maintaining alveolar recruitment; however, optimal PEEP selection in trauma- or postoperative-associated ARDS remains uncertain. Electrical impedance tomography (EIT) enables bedside, real-time assessment of regional ventilation and may support optimal PEEP titration by balancing alveolar overdistension and collapse. This study compares EIT-guided PEEP optimization with the conventional low FiO₂-PEEP strategy in terms of oxygenation and respiratory mechanics in patients with moderate to severe ARDS following trauma or surgery.

DETAILED DESCRIPTION:
This single-center, prospective, randomized controlled trial was designed to evaluate whether EIT-guided PEEP titration improves clinical outcomes in patients with trauma- or postoperative-associated ARDS. Adult intubated patients with moderate to severe ARDS were enrolled.

Patients in the intervention group received PEEP settings guided by electrical impedance tomography, whereas those in the control group were managed according to the lower PEEP/FiO₂ table of the ARDS Network. Other ventilatory parameters and oxygenation targets were set in accordance with ARDS Network recommendations. Supportive care and post-trial PEEP management followed standard ARDS treatment protocols.

The primary outcomes included oxygenation and respiratory mechanics. The secondary outcomes comprised 28-day survival, ventilator-free days at day 28, length of ICU and length of hospital stay, rate of successful ventilator weaning, use of adjunctive therapies (prone positioning, neuromuscular blockade, ECMO), newly developed barotrauma (pneumothorax, pneumomediastinum, and subcutaneous emphysema) excluding cases attributable to invasive procedures) and changes in the SOFA score.

In the intervention group, PEEP was titrated under the guidance of electrical impedance tomography (EIT) according to a protocol:

* Preparation: patients underwent airway suctioning and were deeply sedated (RASS ≤ -3) to abolish spontaneous breathing. PEEP titration was performed using an EIT system (Enlight 2100, Timpel SA, Brazil), with a silicone belt containing 32 surface electrodes positioned at the fourth to fifth intercostal space in accordance with the manufacturer's instructions.
* Pressure-controlled ventilation was applied with an inspiration pressure set at 15 cmH₂O and a set PEEP of 24 cmH₂O, with a maximum airway pressure limit of 40 cmH₂O. Ventilator settings were maintained for 30 seconds with an FiO₂ of 1.0. A decremental PEEP trial was then performed by reducing PEEP in 2 cmH₂O every 30 seconds until a PEEP of 6 cmH₂O was reached or the SpO₂ decreased to ≤ 80%.
* The EIT-guided optimal PEEP was defined as the PEEP level corresponding to the intersection point of the collapse and overdistension curves.

Criteria for discontinuing: PEEP titration was terminated if any of the following occurred: a sustained decrease in mean arterial pressure of > 20 mmHg from baseline, SpO₂ < 88%, or the onset of new cardiac arrhythmias. If the event of discontinuation of the procedure, all ventilator settings were reverted to those applied prior to initiation of the PEEP titration.

In the control group, PEEP was set directly and adjusted according to the lower PEEP/FiO₂ table of the ARDS Network.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated surgical intensive care patients with trauma- or postoperative-associated moderate to severe ARDS, as defined by the 2023 Global Definition of ARDS.

Exclusion Criteria:

* Age <18 or >90 years.
* Severe acute brain injury or acute stroke with Glasgow Coma Scale <8.
* Thoracic trauma with pneumothorax or pneumomediastinum.
* End-stage diseases under palliative care (e.g., metastatic cancer, cirrhosis, end-stage renal disease).
* Severe multiorgan failure with expected survival <7 days.
* Conditions requiring prolonged mechanical ventilation (e.g., Guillain-Barré syndrome, cervical spinal cord injury).
* Contraindications to hypercapnia (e.g., elevated intracranial pressure, acute coronary syndrome).
* Prior use of advanced respiratory therapies (e.g., ECMO, inhaled nitric oxide, prone positioning, high-frequency ventilation).
* Pregnancy, breastfeeding, or skin lesions at electrode placement sites.
* Implanted electrical devices interfering with EIT (e.g., pacemaker, ICD).
* Known allergy to electrode materials.
* Refusal to participate or concurrent enrollment in another study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Oxygenation | at day 0, 1, 2, 3
  PaO₂/FiO₂ ratio
Pulmonary Mechanics | at day 0, 1, 2, 3
  Static Compliance

SECONDARY OUTCOMES:
Ventilator free days | up to 28 days
  Ventilator free days
Length of ICU stay | up to 28 days
  Days of ICU stay
Length of mechanical ventilated days | up to 28 days
  Days of received mechanical ventilation
Barotrauma | up to 28 days
  pneumothorax, pneumomediastinum, and subcutaneous emphysema
Rescue therapies | up to 7 days
  Neuromuscular blocker using, prone postition, ECMO
SOFA | at day 0, 1, 2, 3
  Sequential Organ Failure Assessment
Mortality | up to 28 days
  In-hospital mortality rate

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Anesthesia and Surgical Intensive Care, Viet Duc University Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Costa EL, Borges JB, Melo A, Suarez-Sipmann F, Toufen C Jr, Bohm SH, Amato MB. Bedside estimation of recruitable alveolar collapse and hyperdistension by electrical impedance tomography. Intensive Care Med. 2009 Jun;35(6):1132-7. doi: 10.1007/s00134-009-1447-y. Epub 2009 Mar 3. PMID 19255741
- [Background] Jimenez JV, Weirauch AJ, Culter CA, Choi PJ, Hyzy RC. Electrical Impedance Tomography in Acute Respiratory Distress Syndrome Management. Crit Care Med. 2022 Aug 1;50(8):1210-1223. doi: 10.1097/CCM.0000000000005582. Epub 2022 May 23. PMID 35607967
- [Background] Gao Y, He H, Chi Y, Frerichs I, Long Y, Zhao Z. Electrical impedance tomography guided positive end-expiratory pressure titration in critically ill and surgical adult patients: a systematic review and meta-analysis. BMC Pulm Med. 2024 Nov 23;24(1):582. doi: 10.1186/s12890-024-03394-y. PMID 39580405